CLINICAL TRIAL: NCT00933764
Title: Clinical Performance Evaluation of the Cholestech LDX Cardiac hsCRP Test (CLEAR)
Acronym: CLEAR
Status: Withdrawn | Type: Observational
Sponsor: Abbott RDx Cardiometabolic (Other)
Responsible Party: Meghan Bigelow / Clinical Trial Manager, Inverness Medical Innovations
Other Study IDs: BSTE-0113
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and Serum samples will be retained for reference testing and banking.
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multi-center study designed to assess the accuracy and precision of the Cholestech LDX Cardiac hsCRP test for the quantitative determination of C-reactive protein (CRP) in whole blood, serum and plasma from individuals being assessed for risk of cardiovascular disease. The Cholestech LDX Cardiac hsCRP test consists of the CRP cassette and LDX analyzer and measures CRP with high sensitivity on fingerstick or venous whole blood at the point-of-care (POC). The results of this study are intended to be used for regulatory 510k filings for use as an in vitro diagnostic test.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18 years of age or older) presenting to their physician's office or outpatient clinic for routine or pre-scheduled visits and a candidate for cardiovascular risk assessment.
2. Willing and able to provide written informed consent and comply with study procedures.

Exclusion Criteria:

1. Known hematocrit <30% or > 52%;
2. History of medical conditions - other than risk of cardiovascular disease - that may elevate CRP as listed in Appendix B (e.g., tissue damage, infection, inflammation, malignant neoplasia)
3. Vulnerable populations deemed inappropriate for study by the site's principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals being assessed of their risk of cardiovascular disease. Patients can currently be diagnosed with cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Estimated); Study Completion 2009-11 (Estimated)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - St. Joseph's Research Institute, Atlanta, Georgia
  - Heart and Vascular Research Center of Northern Michigan, Petoskey, Michigan